CLINICAL TRIAL: NCT03543059
Title: A Prospective Observational Study About Adjuvant or Neoadjuvant Chemotherapy Related Adverse Effects in Premenopausal Women With Breast Cancer
Brief Title: A Prospective Observational Study About Adjuvant or Neoadjuvant Chemotherapy Related Adverse Effects in Premenopausal Breast Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, wang shusen, Professor, Sun Yat-sen University
Other Study IDs: SCBCG-021
Record Dates: First submitted 2018-05-21; First posted 2018-06-01 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gonadotropin-Releasing Hormone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- exposure group: exposed to some factors
  Interventions: Drug: GnRH analogue
- control group: not exposed to some factors

INTERVENTIONS:
Drug: GnRH analogue — gonadotrophin releasing hormone analogue
  Groups: exposure group

SUMMARY:
Breast cancer is one of the most common malignant tumor in women. About 60% of breast cancer patients are still in premenopausal status at the time of diagnosis in China. It is a multicenter prospective observational study. We will collect basic information, medical history, chemotherapy-related adverse reactions, and the results of hormone, blood lipid, and bone density test before, during and after adjuvant or neoadjuvant chemotherapy. The aim of the study is to evaluate the effect of chemotherapy on ovarian function and fertility and the protective effect of GnRHa. In addition, the collected information of the subjects are analyzed to provide suggestions for the relevant prevention strategy.

DETAILED DESCRIPTION:
Breast cancer is one of the most common malignant tumor in women, and it occurs at a younger median age in Chinese women than in western white women. About 60% of breast cancer patients are still in premenopausal status at the time of diagnosis in China. Chemotherapy is one of the important treatments for breast cancer, but it brings a series of adverse effects. It is a multicenter prospective observational study. The premenopausal breast cancer women patients who are planning adjuvant or neoadjuvant chemotherapy are enrolled in the study after signing the informed consent form and passing the screening. We collect their basic information, medical history, chemotherapy-related adverse reactions, and the results of hormone, blood lipid, and bone density test before, during and after chemotherapy. The aim of the study is to evaluate the effect of adjuvant or neoadjuvant chemotherapy on ovarian function and fertility and the protective effect of GnRHa by investigating the menopausal symptoms, pregnancy, menstruation condition, hormone levels, blood lipid, bone density, and the usage of GnRHa in the premenopausal women with breast cancer. In addition, the collected information of the subjects are analyzed to provide suggestions for the relevant prevention strategy.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent form has been signed.
2. Breast cancer patients whose age is ≥ 18 years old and have been diagnosed by histological examination.
3. Plan for adjuvant or neoadjuvant chemotherapy

Exclusion Criteria:

1. Postmenopausal women who are defined by any of the following:

   * Previous bilateral oophorectomy;
   * Age ≥ 60 years old;
   * Age <60 years old, menopause at least 12 months, and follicle stimulating hormone [FSH] and estradiol levels in the postmenopausal range.
2. Those who have already received adjuvant or neoadjuvant chemotherapy.
3. Those who have chemotherapy contraindications.
4. Those who have any mental condition that prevents the understanding of the contents of this study and can't provide the complete information required.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Premenopausal women with breast cancer who plan for adjuvant or neoadjuvant chemotherapy
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-06-15 (Estimated); Primary Completion 2021-06-15 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
Pregnancy outcome | 5 years
  The number of patients reporting pregnancy and attempting pregnancy

SECONDARY OUTCOMES:
Rate of ovarian failure | 2 years
  Amenorrhea for 6 months and postmenopausal FSH levels at 24 months (amenorrhea and postmenopausal hormone levels

CONTACTS AND LOCATIONS:
Overall Officials: Shusen Wang, Principal Investigator — Sun Yat-sen University
Locations (1):
- Shusen Wang, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided